CLINICAL TRIAL: NCT04494100
Title: WALANT Technique (Wide Awake Local Anesthesia No Tourniquet) in Association With Analgesic Troncular Blocks at the Wirst for Carpal Tunnel Release.
Brief Title: WALANT Technique (Wide Awake Local Anesthesia No Tourniquet) for Carpal Tunnel Release.
Acronym: WALA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CMC Ambroise Paré (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2020/02
Record Dates: First submitted 2020-07-28; First posted 2020-07-31 (Actual); Last update posted 2021-07-23 (Actual); Status verified 2021-07

CONDITIONS: Carpal Tunnel Release
Keywords: WALANT; Tourniquet; Regional anesthesia; Troncular blocks; Postoperative Analgesia; Ultrasound
MeSH Terms: interventions — Tourniquets; Ropivacaine; Lidocaine; Epinephrine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CONTROL (Active Comparator): Troncular blocks using a long-acting LA + Tourniquet
  Interventions: Procedure: TRONC; Procedure: Tourniquet; Drug: Ropivacaine
- WALANT (Experimental): Troncular blocks using a long-acting LA + WALANT technique using a short-term LA with epinephrine a vasoconstrictor agent
  Interventions: Procedure: TRONC; Procedure: WALANT; Drug: Ropivacaine; Drug: Lidocaine + Epinephrine

INTERVENTIONS:
Procedure: TRONC — injection of 3 to 7 mL of Ropivacaine 3.75 mg/ml per nerve (median and ulnar nerves) and infiltration of 2 ml of Ropivacaine 3.75 mg/ml laterally above the flexion fold of the wrist in order to block the branches of the lateral cutaneous nerve of the forearm, the terminal sensory branch of the musculocutaneous nerve.
Procedure: WALANT — infiltration with 3 to 7 ml of 1% lidocaine (10 mg/ml) combined with 0.005 mg/ml epinephrine and 8.4% sodium bicarbonate in the subcutaneous area in front of the transverse ligament, between the thenar and hypothenar eminences, from the flexion fold of the wrist over a length of 5 cm.
  Arms: WALANT
Procedure: Tourniquet — inflation pressure 75 to 100 mmHg above systolic blood pressure.
  Arms: CONTROL
Drug: Ropivacaine — troncular blocks with Ropivacaine 3.75 mg/ml
Drug: Lidocaine + Epinephrine — WALANT technique with 1% lidocaine (10 mg/ml) combined with 0.005 mg/ml epinephrine
  Arms: WALANT

SUMMARY:
The carpal tunnel release (CTR) is now performed almost exclusively under regional anesthesia (RA) in France. RA requires the use of a pneumatic tourniquet to limit blood flow to the operated extremity and create a bloodless surgical field for a clear visualization of the anatomic structures by the surgeon.

Multiple approaches to block the brachial plexus can be considered. The most common technique is the axillary block (BAX) that provides complete anesthesia for the patient's arm and forearm. This technique offers anesthesia not only for the surgical area but also for the root of the arm where the pneumatic tourniquet is placed. However this technique have limits: the persistence of a motor block in the arm and the forearm that is not compatible with a quick hospital discharge (short term ambulatory hospitalization) and the need for assistance with dressing and eating after surgery. More distal anesthetic techniques are proposed such as the troncular blocks (TRONC) that avoid motor block of the arm and offer an earlier recovery and autonomy for the patient. However, they lead to a poor tolerance to the tourniquet due to its application on a non-anesthetized area.The pain related to the pressure of the tourniquet can occur within the first few minutes of its inflation, get worse over time and persist for several minutes after its deflation. Therefore, TRONC procedure is less often performed compared to the BAX for major surgeries but it remains appropriate for CTR.

The Wide Awake Local Anesthesia No Tourniquet (WALANT) technique is widely used in Canada and has been proposed for hand and wirst minor surgeries. WALANT uses a combination of a local anesthetic (LA) and epinephrine to induce anesthesia and hemostasis in the area of the surgical procedure in order to allow surgeries to be done without the use of tourniquet. Epinephrine is a vasoconstrictor agent that reduces blood flow at surgical site. This bloodless effect is visualized on the skin by a pale color. Thus, WALANT can provide a chemical tourniquet and eliminate the pain from a traditional arm tourniquet. However, this technique is performed with a short-acting LA and does not offer any postoperative analgesia.

The association of TRONC using long-acting LA with the WALANT technique could combine the comfort of a surgery without tourniquet to a long-acting analgesia and thus could provide a superior overall comfort.

The main objective of this prospective, multicentre, randomized, open-label, parallel-group controlled trial is to evaluate the interest of WALANT technique on patient comfort during CTR performed with TRONC, compared to the tourniquet.

DETAILED DESCRIPTION:
This is a multicenter, prospective, randomized, open-label study assessing the interest of the association of the WALANT local infiltration technique with analgesic troncular blocks (TRONC) at the wrist, for the endoscopic CTR.

This study compares two groups:

* CONTROL group (usual technique) : TRONC (using a long-acting LA : Ropivacaine) + Tourniquet
* WALANT group (experimental technique) : TRONC (using a long-acting LA : Ropivacaine) + WALANT ( using a short-term LA : Lidocaine + epinephrine)

RA procedures will be systematically performed under ultrasound guidance, 45 min befor surgery. Before each procedure, a skin disinfection will be carried out using an alcoholic iodine solution. The needle approach will be in-plane (IP) or out-of-plane (OOP). Efficiency will be assessed before transfer to the operating room.

* Troncular blocks (TRONC) Patients will be installed in supine position, the arm at 90° of abduction and in external rotation. The probe will be positioned to have an axial view of the nerves at the wrist. The initial identification of the median (nM) and ulnar (nU) nerves will be systematically done before each TRONC. The nM will be located on the anterior forearm. The nU will be visualized in contact with the ulnar artery in the forearm. The operator will inject 3 to 7 mL of Ropivacaine 3.75 mg/ml per nerve. An infiltration of 2 ml of Ropivacaine 3.75 mg/ml will be performed laterally above the flexion fold of the wrist in order to block the branches of the lateral cutaneous nerve of the forearm, the terminal sensory branch of the musculocutaneous nerve (nMC). A 22 Gauge x 50 mm needle will be used for TRONC.
* WALANT infiltration ("WALANT" group) An infiltration of the subcutaneous area in front of the transverse ligament will be performed between the thenar and hypothenar eminences, from the flexion fold of the wrist over a length of 5 cm. The path of the nM in the palm of the hand will be checked before each procedure. 3 to 7 ml of 1% lidocaine (10 mg/ml) combined with 0.005 mg/ml epinephrine and 8.4% sodium bicarbonate (1 ml per 10 ml of lidocaine) will be injected. The addition of sodium bicarbonate will reduce the pain due to lidocaine injection. A 24 Gauge x 50 mm needle will be used for WALANT.
* Usage of pneumatic Tourniquet A pneumatic tourniquet will be placed at the root of the arm in all patients. A cuff with size and shape adapted to the patient will be used. The tourniquet will be inflated in all patients of "CONTROL" group, and if necessary, corresponding to the failure of the WALANT technique, in patients of "WALANT" group. The inflation pressure will be determined according to the patient's systolic blood pressure (SBP). It will be inflated 75 to 100 mmHg above SBP

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing endoscopic carpal tunnel release
* Consent for participation
* Affiliation to a social security system

Exclusion Criteria:

* Chronic pain syndrome or fibromyalgia
* Contraindication for locoregional anesthesia
* ASA 4
* Pregnant or breastfeeding women
* Patients under protection of the adults(guardianship, curators or safeguard of justice)
* Communication difficulties or neuropsychiatric disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-09-11 (Actual); Primary Completion 2021-06-25 (Actual); Study Completion 2021-07-05 (Actual)

PRIMARY OUTCOMES:
Patient comfort during CTR | 4 hours
  Pain score using a Visual Analogue Sclae (VAS) ranging from 0 to 10 (0= completely painless, 10= extremely painfull).

SECONDARY OUTCOMES:
Quality of the endoscopic surgical procedure | 4 hours
  Numeric Rating Scale (NRS) for visualization during endoscopic surgery ranging from 0 to 5 ( 0=very poor conditions; 5=optimal conditions)
Troncular block success | 30 minutes
  Sensory perception to pin-prick on the specific territories of the median, ulnar and radial nerves at 10, 20 and 30 minutes post injection using a 3-point rating: 0 = absence of block (sharp sensation to pinprick), 1 = analgesia (dull sensation to pinprick), 2 = anesthesia (loss of sensation to pinprick)The need for an additional block, an intraoperative surgical infiltration or a sedation will be noted.
WALANT technique success | 30 minutes
  Modification (or not) of the skin color near the injection area at 10, 20 and 30 minutes postinjection.
Hemostasis quality for the WALANT group | 4 hours
  Usage (or not) of tourniquet.
Patient satisfaction | 4 hours
  Patient satisfaction score collected in post-anesthesia care unit (PACU) using a Numeric Rating Scale (NRS-Satisfaction) ranging from 0 (very unsatisfied) to 10 (very satisfied).
Surgery duration | 4 hours
  Time (in minutes) between the skin incision and the last suture.
Rate of complications | 20 days
  Incidence of complications related to RA procedure

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Clinique Jouvenet, Paris, Île-de-France Region
  - Clinique Rémusat, Paris, Île-de-France Region

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bloc S, Squara P, Quemeneur C, Doirado M, Thomsen L, Merzoug M, Naudin C, Le Sache F. Wide Awake Local Anesthesia No Tourniquet (WALANT) technique improves the efficiency of distal nerve blocks for carpal tunnel release. Anaesth Crit Care Pain Med. 2023 Aug;42(4):101229. doi: 10.1016/j.accpm.2023.101229. Epub 2023 Apr 7. PMID 37031817